CLINICAL TRIAL: NCT04315688
Title: A Prospective Non-interventional Study Investigating the Treatment Effect of Tresiba® in Adult Patients With Type 2 Diabetes in Russia
Brief Title: A Research Study, Looking at How Tresiba® Works in People With Type 2 Diabetes in Local Clinical Practice in Russia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4589; U1111-1236-4887 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tresiba®: Patients with type 2 diabetes
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Treatment with Tresiba® with or without anti-diabetes medication (as per local label), as prescribed by the participant's physician. The study population will include adult patients with type 2 diabetes, both insulin naïve and previously insulin treated, for whom the treating physician has decided to initiate treatment with Tresiba®, independent of the decision to include the patient in the study.

SUMMARY:
The purpose of the study is to collect information on how Tresiba® works in real world patients with Diabetes Mellitus, Type 2 (type 2 diabetes). Participants will get Tresiba® as prescribed by their doctor. The study will last for around 6 to 8 months. Participants will be asked questions about their health and their diabetes treatment as part of their normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Tresiba® has been made by the patient and the treating physician before and independently from the decision to include the patient in this study.
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes and treated with any antihyperglycemic medication(s), except Tresiba® (insulin degludec), for at least 26 weeks prior to Informed consent and Initiation Visit (Visit 1).
* Available and documented HbA1c value 12 weeks or less prior to initiation of Tresiba® treatment.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Hypersensitivity to the active substance or to any of the excipients as specified in the Tresiba® local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change in laboratory measured glycated haemoglobin (HbA1c) (% point) | From baseline (week -12 to 0) to end of study (week 26-36)
  % point
Change in laboratory measured HbA1c (mmol/mol) | From baseline (week -12 to 0) to end of study (week 26-36)
  mmol/mol

SECONDARY OUTCOMES:
Change in laboratory measured fasting plasma glucose (FPG) | From baseline (week -12 to 0) to end of study (week 26-36)
  mg/dL
Change in laboratory measured FPG | From baseline (week -12 to 0) to end of study (week 26-36)
  mmol/L
Change in daily insulin doses (basal insulin) | From baseline (week -12 to 0) to end of study (week 26-36)
  units/day
Change in daily insulin doses (prandial insulin) | From baseline (week -12 to 0) to end of study (week 26-36)
  units/day
Change in daily insulin doses (total insulin) | From baseline (week -12 to 0) to end of study (week 26-36)
  units/day
Change in number of patient reported overall non-severe hypoglycaemic episodes | Pre and Post- initiation of treatment with Tresiba®. Episodes occurring within 4 weeks prior to initiation of treatment with Tresiba® (week -12 to 0) and within 4 weeks prior to end of study (week 26 to 36)
  Number of episodes
Change in number of patient reported nocturnal non-severe hypoglycaemic episodes | Pre and Post- initiation of treatment with Tresiba®. Episodes occurring within 4 weeks prior to initiation of treatment with Tresiba® (week -12 to 0) and within 4 weeks prior to end of study (week 26 to 36)
  Number of episodes
Change in number of patient reported severe hypoglycaemic episodes (overall) | Pre and Post- initiation of treatment with Tresiba®. Episodes occurring within 4 weeks prior to initiation of treatment with Tresiba® (week -12 to 0) and within 4 weeks prior to end of study (week 26 to 36)
  Number of episodes
Reason(s) for discontinuing treatment with Tresiba® during the treatment period, if applicable (according to pre-specified response options) | After initiation of treatment with Tresiba® (week 0) until treatment discontinuation (week 26-36)
  Number of participants per response option

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (33):
- Russia (33):
  - Novo Nordisk Investigational Site, Alushta
  - Novo Nordisk Investigational Site, Belogorsk
  - Novo Nordisk Investigational Site, Bryansk
  - Novo Nordisk Investigational Site, Chapayevsk
  - Novo Nordisk Investigational Site, Chelyabinsk
  - Novo Nordisk Investigational Site, Dyurtyuli
  - Novo Nordisk Investigational Site, Elista
  - Novo Nordisk Investigational Site, Ivanovo
  - Novo Nordisk Investigational Site, Kaluga
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Krasnodar
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Lipetsk
  - Novo Nordisk Investigational Site, Lyskovo
  - Novo Nordisk Investigational Site, Magnitogorsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Moscow Region, Dolgoprudny
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Odintsovo, Moscow Region
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Rostov-on-Don
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Peterburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Sergiyev Posad
  - Novo Nordisk Investigational Site, Sevastopol’
  - Novo Nordisk Investigational Site, Sovetskiy
  - Novo Nordisk Investigational Site, Syktyvkar
  - Novo Nordisk Investigational Site, Tula
  - Novo Nordisk Investigational Site, Ufa
  - Novo Nordisk Investigational Site, Voskresensk
  - Novo Nordisk Investigational Site, Vyksa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com